CLINICAL TRIAL: NCT01174511
Title: Clinical Trial Study for Evaluation of A-1 Cool Cream Efficacy for Treatment Patients With Atopic Dermatitis
Brief Title: Evaluation of A-1 Cool Cream Efficacy for Treatment Atopic Dermatitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Prof. Arieh Ingber - Head of Department of Dermatology and Venereology - Hadassah Medical Center, Hadassah Medical Organization, Jerusalem, Israel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 0124-10-HMO-ctil
Record Dates: First submitted 2010-08-02; First posted 2010-08-03 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2010-07

CONDITIONS: ATOPIC DERMATITIS
Keywords: ATOPIC DERMATITIS; A-1 COOL CREAM
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A-1 COOL cream (Experimental): A research product - A-1 COOL cream contain herbal medicine plants basically :
  1. WATER PETROLATUM
  2. WILD YAM (DIOSCOREA VILLOSA) EXTRACT
  3. SORBITAN SESQUIOLEATE
  4. CALENDULA OFFICINALIS EXTRACT
  5. MINERAL OIL
  6. ARNICA MONTANA EXTRACT
  7. MICROCRYSTALLINE WAX
  8. LICORICE (GLYCYRRHIZA GLABRA) EXTRACT
  9. DECYL OLEATE
  10. DICOCOYL PENTAERYTHRITYL DISTEARYL CITRATE
  11. BEESWAX
  12. ALUMINUM STEARATES
  Interventions: Drug: A -1 Cool Cream,Vaselin ointment
- Vaselin ointment (Placebo Comparator): Using the study as placebo.
  Interventions: Drug: A -1 Cool Cream,Vaselin ointment

INTERVENTIONS:
Drug: A -1 Cool Cream,Vaselin ointment — A- 1 Cool Cream applied to flexural aspects of the upper and lower limb on the one site of patient and placebo (Vaseline ointment) applied to other site of the upper and lower limb in the itch patient. Applying the ointment will be a regular time, twice a day for 5 consecutive days

SUMMARY:
Atopic dermatitis (AD) is a chronic inflammatory skin disease, affecting 20% of all babies and children around the world. Diagnosis of atopic dermatitis is clinical and depends on the existence of at least two out of the four following criteria: itching, a chronic disease course with exacerbations and remission ,rash with characteristic distribution and shape , atopia of the patient or family by history.

Initial treatment is based on keeping skin moist and avoiding a flare-provoking stimuli and allergens. The research product A-1 COOL is a skin cream approved by the Israeli Ministry of Health for cooling down of skin irritation. A-1 COOL is rich in herbal medicine ingredients and does not contain steroids.A-1 COOL can be beneficial in Atopic Dermatitis patients due to its following action mechanisms: sealing of the inflamed skin and retention of water, prevention of the itching cycle by keeping the skin moist, disinfection of the skin by the herbal ingredients.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a chronic inflammatory skin disease, affecting 20% of all babies and children around the world. In 90% of the cases the disease first appears before the age of five and in 65% of the cases it is already apparent at infancy but it may occur at any age.

Diagnosis of atopic dermatitis is clinical and depends on the existence of at least two out of the four following criteria: itching, a chronic disease course with exacerbations and remission ,rash with characteristic distribution and shape , atopia of the patient or family by history.

Initial treatment is based on keeping skin moist and avoiding a flare-provoking stimuli and allergens. Topical ointments which grease the skin have shown and reduction of skin inflammation. These products can include active substances such as steroids and anti-inflammatory compounds.

Systemic treatments for atopic dermatitis mainly include steroids and cyclosporine.

The research product A-1 COOL is a skin cream approved by the Israeli Ministry of Health for cooling down of skin irritation. A-1 COOL is rich in herbal medicine ingredients and does not contain steroids.A-1 COOL can be beneficial in Atopic Dermatitis patients due to its following action mechanisms: sealing of the inflamed skin and retention of water, prevention of the itching cycle by keeping the skin moist, disinfection of the skin by the herbal ingredients.

ELIGIBILITY:
Inclusion Criteria:

* patient with atopic dermatitis,
* Hebrew-speaking men and women,
* over 18 years old.

Exclusion Criteria:

* hospital where the diagnosis of atopic dermatitis is not sure,
* patients under the age of 18, pregnant women, no - helpless, soldiers and prisoners,
* patients with atopic dermatitis treated with systemic preparations such as cyclosporine, steroids, antibiotics, methotrexate, biological preparations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of A-1 cool treatment by TIS score | 5 DAYS
  Initially, we will evaluate the disease severity in all the research subjects by SCORAD SCORE and TIS score.Thereafter we will apply to each subject's flexor aspects of the upper or lower limbs on one side the research product and on the other the placebo.This treatment will be given twice a day at specific times for 5 days. As ameasure to evaluate the efficacy of A-1 COOL treatment wiil be use the Three- item severity score (TIS)- reviewer redness, edema ,scratch marks.Severity of these symptoms wiil be evaluated from 0 to 3 points scale.

REFERENCES:
- See also: Katoh N.Future perspectives in the treatment of atopic dermatitis. — http://www.ncbi.nlm.nih.gov/pubmed/19583684